CLINICAL TRIAL: NCT02974140
Title: A Prospective, Multicenter, Randomized Evaluation of Refractive Predictability in Patients With or Without Corneal Astigmatism (Maximum Allowable up to 1.25D) When Using the Cataract Refractive Suite and Standard Manual Techniques
Brief Title: Cataract Refractive Suite Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Management Decision
Sponsor: Alcon, a Novartis Company (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTK246-P001
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-08

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- CRS (Experimental): First surgical eye randomized to Cataract Refractive Suite with second surgical eye (fellow eye) assigned to standard manual technique. Second eye surgery conducted within 7-14 days of the first eye surgery.
  Interventions: Device: Cataract Refractive Suite (CRS); Procedure: Standard manual technique
- Manual (Active Comparator): First surgical eye randomized to standard manual technique with second surgical eye (fellow eye) assigned to Cataract Refractive Suite. Second eye surgery conducted within 7-14 days of the first eye surgery.
  Interventions: Device: Cataract Refractive Suite (CRS); Procedure: Standard manual technique

INTERVENTIONS:
Device: Cataract Refractive Suite (CRS) — Configuration consisting of Verion™ Image Guided System, LenSx® Laser and ORA™ System with VerifEye+™ (with or without VerifEye Lynk), combined for use in surgical pre-op planning and during cataract surgery
Procedure: Standard manual technique — Standard biometry for intra-ocular lens (IOL) calculation and cataract removal using phacoemulsification technique

SUMMARY:
The purpose of this study is to compare the refractive predictability (prediction error) between the Cataract Refractive Suite (CRS) and standard manual technique at one month post-operative

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with bilateral cataracts;
* Planned cataract surgery and implantation of ReSTOR +2.5 D multifocal intraocular lens (IOL) in both eyes;
* Clear intraocular media, other than cataract, in study eye(s);
* Willing and able to complete all required postoperative visits;
* Able to comprehend and sign a statement of informed consent;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Significant irregular corneal astigmatism;
* History of or current severe dry eyes, retinal/uveal pathology or concurrent ocular disease;
* Previous intraocular or corneal refractive surgery, corneal transplant, or retinal detachment;
* Any inflammation or edema (swelling) of the cornea;
* Pregnant;
* Other protocol-specified exclusion criteria may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2017-07-25 (Actual); Study Completion 2017-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Manager, GCRA, Study Director — Alcon, A Novartis Division
Locations (3):
- United States (3):
  - Alcon Investigative Site, Panama City, Florida
  - Alcon Investigative Site, Stillwater, Minnesota
  - Alcon Investigative Site, Hurst, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 3 investigative sites located in the United States.
Pre-assignment Details: This reporting group includes all enrolled subjects (39).
Units Other Than Participants: eyes
Groups:
- All Study Subjects: Cataract extraction surgery with either Cataract Refractive Suite (CRS) or manual technique in the study eye, defined as the eye with the worst preoperative corrected distance visual acuity (CDVA), with the alternate procedure in the fellow eye
Period: Overall Study
Arm/Group | All Study Subjects
Started | 39; 78 eyes
CRS (Left or Right Eye) (Cataract surgery using Cataract Refractive Suite, as randomized) | 38; 38 eyes
Manual (Fellow Eye) (Cataract surgery using standard manual technique) | 38; 38 eyes
Completed | 0; 0 eyes
Not Completed | 39; 78 eyes
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 1
Not completed — Study Terminated by Sponsor | 36

BASELINE CHARACTERISTICS:
Population: This analysis population includes all eyes that were randomized and for which an intraocular lens (IOL) was successfully implanted (Full Analysis Set).
Groups:
- All Study Subjects: Cataract extraction surgery with either CRS or manual technique in the study eye, defined as the eye with the worst preoperative corrected distance visual acuity (CDVA), with the alternate procedure in the fellow eye
Arm/Group | All Study Subjects
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 38
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Manifest Refraction Spherical Equivalent (MRSE) Within 0.5 Diopter (D) of Predicted Postoperative Spherical Equivalent at Month 1
Description: Manifest refraction spherical equivalent (MRSE) was calculated as follows: sphere + 1/2 cylinder. The sphere and cylinder values were from the manifest refraction assessment. Manifest refraction was assessed at 4 meters under photopic lighting conditions using a phoropter. Due to early termination of the study and limited sample size, a statistical inference test was not carried out as planned.
Time Frame: Day 20-40 from second implantation
Population: Full Analysis Set with data available
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Groups:
- Suite: Cataract surgery using Cataract Refractive Suite
- Manual: Cataract surgery using standard manual technique
Arm/Group | Suite | Manual
Number analyzed (Participants) | 36 | 36
Number analyzed (Eyes) | 36 | 36
percentage of eyes | 80.6 | 69.4

2. Secondary Outcome: Cumulative Dissipated Energy (CDE)
Description: Cumulative Dissipated Energy (CDE) represents the energy dissipated of the ultrasound tip and infusion sleeve at the incision point during the removal of cataractous lens. CDE was reported on the Vision System interface and measured in percent-seconds. A lower CDE indicates that less energy was expended in the eye. Due to early termination of the study and limited sample size, a statistical inference test was not carried out as planned.
Time Frame: Day 0 (operative day), each eye
Population: Full Analysis Set with data available
Measure: Mean (Standard Deviation); unit: percent-seconds
Units Other Than Participants: Eyes
Arm/Group | Suite | Manual
Number analyzed (Participants) | 37 | 38
Number analyzed (Eyes) | 37 | 38
percent-seconds | 3.396 (2.4620) | 4.032 (2.6022)

3. Secondary Outcome: Estimated Aspiration Fluid Used During Surgery
Description: Aspiration fluid (amount of fluid used during the removal of the cataractous lens) was measured in milliliters (ml). A lower value indicates less fluid used during the procedure. Due to early termination of the study and limited sample size, a statistical inference test was not carried out as planned.
Time Frame: Day 0 (operative day), each eye
Population: Full Analysis Set with data available
Measure: Mean (Standard Deviation); unit: ml
Units Other Than Participants: Eyes
Arm/Group | Suite | Manual
Number analyzed (Participants) | 37 | 38
Number analyzed (Eyes) | 37 | 38
ml | 58.6 (16.48) | 54.0 (11.57)

4. Secondary Outcome: Phaco Aspiration Time Spent During Surgery
Description: Phaco aspiration time (the average time the surgeon took to complete the phacoemulsification) was measured in seconds. A lower value indicates that the surgeon spent less time aspirating fluid and material from the eye during surgery. Due to early termination of the study and limited sample size, a statistical inference test was not carried out as planned.
Time Frame: Day 0 (operative day), each eye
Population: Full Analysis Set with available data
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Eyes
Arm/Group | Suite | Manual
Number analyzed (Participants) | 37 | 38
Number analyzed (Eyes) | 37 | 38
seconds | 197.9 (77.06) | 173.3 (57.89)

ADVERSE EVENTS:
Time Frame: Surgery through study completion, an average of 1 month.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users, or other persons, whether or not related to the investigational medical device. AEs were obtained through solicited and spontaneous comments from subjects and observations by the Investigator. "At risk" population for ocular AEs is reported in units of eyes. Two subjects had only 1 eye treated (39 overall subjects, 38 eyes in each group).
Groups:
- Suite (Ocular): Eyes for which the LenSx was activated and a laser cut was initiated
- Manual (Ocular): Eyes for which the incision was initiated using standard manual techniques
- Nonocular: Subjects for which cataract surgery was conducted in one or both eyes
Arm/Group | Suite (Ocular) | Manual (Ocular) | Nonocular
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38 | 0/39
Serious Adverse Events (participants affected / at risk) | 1/38 | 0/38 | 0/39
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Suite (Ocular) (N=38) | Manual (Ocular) (N=38) | Nonocular (N=39)
Retinal Tear (Eye disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT02974140/SAP_000.pdf
  • Study Protocol (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT02974140/Prot_001.pdf